CLINICAL TRIAL: NCT00956046
Title: Immunogenicity and Safety of Multiple Formulations of an Intramuscular Inactivated, Split Virion Swine-origin A/H1N1 Influenza Vaccine With and Without Adjuvant in Healthy European Subjects Aged 6 to 35 Months
Brief Title: A Study of Swine-origin A/H1N1 Influenza Vaccines in Healthy Europeans Children Aged 6 to 35 Months
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GPF09; UTN: U1111-1111-5029 (Other: WHO); 2009-013858-32 (EudraCT Number)
Record Dates: First submitted 2009-08-03; First posted 2009-08-11 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Influenza; Swine-origin A/H1N1 Influenza
Keywords: Influenza; Pandemic Flu; Swine-origin A/H1N1 Influenza; Swine-origin Influenza Virus; Infants
MeSH Terms: conditions — Influenza, Human | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A/H1N1 Vaccine Group 1 (Experimental): All participants will receive A/H1N1 Influenza vaccine formulation 1 at Visits 1 and 2; and a subset will receive a trivalent influenza vaccine (TIV) at Month 13 (antibody persistence subset)
  Interventions: Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated)
- A/H1N1 Vaccine Group 2 (Experimental): All participants will receive A/H1N1 Influenza vaccine formulation 2 at Visits 1 and 2; and a subset will receive a trivalent influenza vaccine (TIV) at Month 13 (antibody persistence subset).
  Interventions: Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated + Adjuvant)
- A/H1N1 Vaccine Group 3 (Experimental): Participants will receive A/H1N1 Influenza vaccine formulation 3
  Interventions: Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated + adjuvant)

INTERVENTIONS:
Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated) — 0.5 mL, Intramuscular on Day 0 and Day 21 (all participants); and 0.5 mL of a trivalent influenza vaccine (TIV) at Month 13 (antibody persistence subset).
  Arms: A/H1N1 Vaccine Group 1
Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated + Adjuvant) — 0.5 mL, Intramuscular on Day 0 and Day 21 (all participants); and 0.5 mL of a trivalent influenza vaccine (TIV) at Month 13 (antibody persistence subset)
  Arms: A/H1N1 Vaccine Group 2
Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated + adjuvant) — 0.5 mL, Intramuscular on Day 0 and Day 21
  Arms: A/H1N1 Vaccine Group 3

SUMMARY:
The purpose of this study is to generate data on immunogenicity and safety of the monovalent H1N1 vaccine in support of the development and registration.

Primary objectives:

* To describe the immune response to vaccines 21 days after each vaccination in all participants.
* To describe the antibody persistence eight months after the first vaccine administration using hemagglutination inhibition (HAI) method in a subset of participants who received two half-doses of either formulation 1 or 2.
* To describe the immune response against the A/H1N1 strain using the HAI method 21 days after last vaccination with the 2010-2011 NH seasonal Trivalent Influenza Vaccine (TIV) administered 13 months after the first vaccination in a subset of subjects who received two half-doses of either t either formulation 1 or 2 of the A/H1N1 influenza vaccines as primary series.
* To describe the safety profile of each vaccine in all participants.

DETAILED DESCRIPTION:
All participants will receive two injections of their randomized vaccine on Day 0 and Day 21, respectively.

A subset of the participants eligible who received two half-doses of either formulation 1 or 2 will also be proposed to receive the 2010-2011 Northern Hemisphere (NH) seasonal Trivalent Influenza Vaccine (TIV) 13 months after the first vaccination as Follows:

* Subjects less than 36 months at the time of TIV injection will receive two half-doses and additional sampling for immunogenicity assessment (one before the first TIV vaccination and one 21 days after last TIV vaccination).
* Subjects aged more than 36 months at the time of TIV injection will receive a full TIV dose and additional sampling for immunogenicity assessment (one before TIV vaccination and one 21 days after TIV vaccination).

ELIGIBILITY:
Inclusion Criteria :

All subjects

* Aged 6 to 35 months on the day of inclusion
* Informed consent form has been signed and dated by the parent(s) or other legally acceptable representative
* Subject and parent/legal representative are able to attend all scheduled visits and to comply with all trial procedures
* Completion of vaccination according to the national immunization schedule.

Subjects ≥ 6 to < 24 months of age - Born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg

At Month 8 for antibody persistence assessment:

* Having received two half-doses of either the formulation 1 or 2 of the vaccine
* Addendum 1 to Informed Consent Form has been signed and dated by the parents or other legally acceptable representative.

At Visit 06, for subjects eligible for the Antibody persistence evaluation who will receive the Trivalent Influenza Vaccine (TIV):

- Addendum 2 to Informed Consent Form has been signed by the subject's parents/legal representative.

Exclusion Criteria :

All subjects

* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination
* Planned receipt of any vaccine prior to the Day 42 blood sample
* Receipt of blood or blood-derived products in the past 3 months which might interfere with the assessment of immune response
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B antigen, or Hepatitis C as reported by parents/legal representative
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances
* Thrombocytopenia contraindicating intramuscular (IM) vaccination as reported by parents/legal representative
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion contraindicating IM vaccination
* Chronic illness that in the opinion of the Investigator is at a stage where it might interfere with trial conduct or completion
* Family members of the employees or the Investigator
* Previous participation in a trial investigating a vaccine with the swine-origin A/H1N1 influenza strain
* Confirmed infection with the swine-origin A/H1N1 influenza strain (different from the seasonal strain) in 2009
* Febrile illness (temperature ≥ 38.0°C) or moderate or severe acute illness/infection on the day of vaccination, according to Investigator judgment
* Receipt of any allergy shots and/or seasonal allergy medication in the 7-day period prior to enrollment (vaccination), or scheduled to receive any allergy shots and/or seasonal allergy medication in the 7-day period after enrollment (vaccination)

Subjects ≥ 6 to < 24 months of age - History of seizures

At Month 8, for antibody persistence assessment:

- Subjects who received, in the context of a pandemic immunization program, another A/H1N1 pandemic influenza vaccine than the Investigational Medicinal Products.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 401 (Actual)
Dates: Start 2009-09; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: To provide information concerning the immunogenicity of Swine A/H1N1 influenza vaccines | 21 days post vaccination
Safety: To provide information concerning the safety in terms of solicited injection site and systemic reactions of Swine A/H1N1 influenza vaccines. | 0-7 days post-vaccination and entire study duration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (13):
- Finland (13):
  - Espoo
  - Helsinki
  - Jarvenpaa
  - Kokkola
  - Kotka
  - Kuopio
  - Lahti
  - Oulu
  - Pori
  - Seinäjoki
  - Tampere
  - Turku
  - Vantaa

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com